CLINICAL TRIAL: NCT00715416
Title: Balloon Angioplasty vs. Primary Stenting of Femoropopliteal Arteries Using Self-Expandable Nitinol Stents - a Randomized Controlled Trial
Brief Title: PTA vs. Primary Stenting of SFA Using Self-Expandable Nitinol Stents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vienna General Hospital (Other)
Responsible Party: Prof. Martin Schillinger, General Hospital of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1/2006
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2006-01

CONDITIONS: Peripheral Vascular Diseases; Intermittent Claudication; Angioplasty
Keywords: peripheral vascular diseases; Intermittent Claudication; Angioplasty
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): primary nitinol stent placement of superficial femoral artery lesions
  Interventions: Device: Nitinol stent; Procedure: Nitinol Stent Placement
- 2 (Active Comparator): balloon angioplasty of superficial artery lesions with secondary stent placement in case of >30% residual stenosis after the procedure
  Interventions: Device: Nitinol stent

INTERVENTIONS:
Device: Nitinol stent — Interventions are performed percutaneously from either an antegrade or an over-the-bifurcation approach. After insertion of an 6 French sheath, 5000 IU of heparin are administered intra-arterially. After passage of the stenosis/occlusion with the guide wire, patients are randomized to either PTA or primary stent implantation. For standardized documentation of the lesion morphology and comparability during follow-up, a ruler is fixed at the patients thigh with the distal end exactly overlapping at the upper edge of the patella. As a bail-out procedure in the PTA group, stent placement is performed in cases with a residual stenosis of more than 30% in the worst view angiogram.
Procedure: Nitinol Stent Placement — Balloon angioplasty compared to primary stent implantation for long segment superficial femoral artery lesions
  Other Names: Product: peripheral stent system; Type: ASTRON; EC class: IIb; Certificate number: G1 01 10 10275 193; EC number: 0123; Date of issue: 26.10.2001
  Arms: 1

SUMMARY:
The investigators evaluated whether primary implantation of a self-expanding nitinol stent yielded anatomical and clinical benefits superior to those afforded by percutaneous transluminal angioplasty with optional secondary stenting.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic peripheral artery disease with severe intermittent claudication (Fontaine stage IIb)
* critical limb ischemia in patients with stenosis or occlusions originating in the SFA
* up to 25 cm length of stenosis/occlusion

Exclusion Criteria:

* previous bypass surgery at the site of treatment
* history of intolerance of anti-platelet therapy
* adverse reaction to heparin
* bleeding diathesis
* creatinine >2.5 mg/dL
* active bacterial infection
* allergy to contrast media
* previous stent placement at or immediately adjacent to the target lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
occurrence of a >50% restenosis at the treated segment at 6 months postintervention as determined by CTA (in-segment restenosis). | 3, 6, 12 months

SECONDARY OUTCOMES:
ultrasound patency, clinical patency, target vessel and target lesion revascularization, cardiovascular events, quality of life at 3, 6 and 12 months after the procedure | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schilliger, Prof, Principal Investigator — General Hospital of Vienna, Department of Angiology; Martin Schillinger, Prof, Principal Investigator — General Hospital of Vienna
Locations (1):
- University Hospital of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699